CLINICAL TRIAL: NCT02466334
Title: CGRP's Cluster Headache Inducing Abilities in Cluster Headache Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Song Guo, Medical doctor, Ph.d. student, Danish Headache Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: H-15006836
Record Dates: First submitted 2015-05-21; First posted 2015-06-09 (Estimated); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Cluster Headache
MeSH Terms: conditions — Cluster Headache | interventions — Calcitonin; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active (Active Comparator): 1.5µg/min IV calcitonin-gene related peptide for 20 minutes
  Interventions: Drug: Calcitonin-Gene Related Peptide
- Placebo (Placebo Comparator): IV placebo for 20 minutes
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Calcitonin-Gene Related Peptide — 1,5 µg/min of IV CGRP over 20 mins
  Other Names: CGRP
  Arms: Active
Drug: Placebo — 40 ml of normal saline over 20 mins
  Other Names: Normal saline
  Arms: Placebo

SUMMARY:
It has previously been shown that nitroglycerine induces cluster headache attacks in episodic cluster headache patients (ECH patients) in bouts but not in remission phase. Furthermore, plasma concentrations of calcitonin gene-related peptide (CGRP) have been shown to be significantly higher during, but not before and after, an attack.

The attack appears around 20-40 min after nitroglycerine infusion with vasodilatation. During this latency period preceding the attack, no increase in CGRP plasma concentrations is seen. CGRP induces migraine attacks in 65% of migraine patients, and CGRP antagonists as well as monoclonal antibodies against CGRP are effective in migraine treatment.

Based on the above the investigators hypothesize the following:

1. Provoking ECH patients in bout with CGRP triggers cluster headache attacks
2. Provoking ECH patients in remission with CGRP does not trigger cluster headache attacks
3. Provoking chronic cluster headache patients with CGRP triggers cluster headache attacks more often than in ECH patients.

ELIGIBILITY:
Inclusion Criteria:

* Fulfillment of IHS criteria for cluster headache either chronic or episodic
* Patients in bouts 1-32 attacks per week
* Patients in remission minimum of 1 month remission time
* fertile women must use safe contraception

Exclusion Criteria:

* All other primary types of headache
* headache 8 hours or less before study day begins
* pregnant or lactating women
* any history or clinical sigs of hyper/hypotension, heart disease, mental disorder, substance abuse, or other illness deemed relevant by the medical doctor assessing the patient

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2015-06; Primary Completion 2017-03 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Differences in occurence of cluster headache attacks on CGRP day compared to placebo day in all three groups | 90 min after administration of study drug
  Occurence of experimentally induced cluster headache attack yes/no
AUC headache on CGRP day compared to placebo day in all three groups | 90 min after administration of study drug
  Using 90 min headache questionnaire
Time to maximum headache score on CGRP day compared to placebo day in all three | 90 min after administration of study drug
  Using 90 min headache questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Messoud Ashina, MD, PhD,DMSc, Principal Investigator — Danish Headache Center
Locations (1):
- Danish Headache Center, Copenhagen, Glostrup, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Vollesen ALH, Snoer A, Beske RP, Guo S, Hoffmann J, Jensen RH, Ashina M. Effect of Infusion of Calcitonin Gene-Related Peptide on Cluster Headache Attacks: A Randomized Clinical Trial. JAMA Neurol. 2018 Oct 1;75(10):1187-1197. doi: 10.1001/jamaneurol.2018.1675. PMID 29987329